CLINICAL TRIAL: NCT03436966
Title: Role Of Computed Tomography Enterography in Diagnosis of Inflammatory Bowel Disease
Brief Title: Role of Multislice CT in Diagnosis of Inflammatory Bowel Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Heba Abo Elmakarem Ahmed, Principle investigator, Assiut University
Other Study IDs: MSCT in IBD
Record Dates: First submitted 2018-02-13; First posted 2018-02-19 (Actual); Last update posted 2018-02-20 (Actual); Status verified 2018-02

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: MULTI SLICE CT — Positive enteric contrast, can, however, obscure IV contrast enhancement of the bowel wall. In addition, positive oral contrast agents opacify but do not always well distend the bowel. IV contrast is administered and images are acquired in the portal venous phase, which is optimized for visceral organ evaluation.

SUMMARY:
Aim of the work: To evaluate the role of CT in diagnosis of IBD

DETAILED DESCRIPTION:
Inflammatory bowel disease (IBD): is a chronic idiopathic disease affecting the gastrointestinal (GI) tract that is comprised of two separate, but related intestinal disorders; Crohn s disease (CD) and ulcerative colitis (UC), IBD is thought to result from an exaggerated and inappropriate immune response to gut luminal microbes in genetically, susceptible individuals who are exposed to environmental risk factors. IBD is most common in North America and western and northern Europe, where incidence rates for UC and CD range from 2.2-24.3 per 100000 person years, It is estimated that more than 1.4 million Americans and as many as 2.5-3 million, Europeans have IBD. While UC and CD share some features, the diseases are distinct. Perhaps the most important differences are that while the chronic inflammation seen in UC is limited to the large intestine and affects only the intestinal mucosa, the inflammation in CD can occur at any location(s) along the GI tract and is often transmural, predisposing patients with CD to the development of penetrating (fistulizing) and fibro stenotic (stricturing) phenotypes that are not typically seen in UC. In some cases, UC and CD are not distinguishable and a diagnosis of IBD unclassified (IBD-U) is made although clinical features of IBD-U tend to mirror those of UC Clinical manifestations of UC include diarrhea, with or without blood, abdominal pain, tenesmus, and fecal urgency, while the manifestations of CD are more variable depending on the extent and location of the GI inflammation. CD with predominantly colonic involvement often presents in similar fashion to UC whereas in small bowel CD, diarrhea and rectal bleeding are seen less frequently and symptoms, fever, fatigue and weight loss are common.

ELIGIBILITY:
Inclusion Criteria:

* Patient in the age group between 15&40 and another age group between 50&80 with inflammatory bowel disease.

Exclusion Criteria:

* Patients with any general contraindication to Radiation of CT especially pregnant women.
* Patients with any general contraindication to contrast, impaired renal function & hypersensitivity.
* Patients of the age group below 15 years old.

Ages: 15 Years to 80 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: * Number of 30 Patients with inflammatory bowel disease will be included in the study.
  * CT scans are typically performed for IBD evaluation following administration of both oral and IV contrast to detect bowel wall abnormalities and abnormal enhancement[6]
  * Conventional CT uses positive enteral contrast agents, usually water soluble containing solutions, which increase the attenuation of the bowel lumen and of bowel wall abnormalities and extraluminal fluid collections.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2018-10 (Estimated); Primary Completion 2019-09 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of inflammatory bowel disease by MSCT enterography | baseline
  detect the early complication of the disease: fistula, stricture, fibofatty changes by enterography

CONTACTS AND LOCATIONS:
Overall Officials: shreef abd, prof, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Loftus EV Jr. Clinical epidemiology of inflammatory bowel disease: Incidence, prevalence, and environmental influences. Gastroenterology. 2004 May;126(6):1504-17. doi: 10.1053/j.gastro.2004.01.063. PMID 15168363